## (OCTOBER-4: INFORMED VOLUNTARY ACTION FORM (INTERVENTION GROUP)

#### **Dear Participant**

# **Description of The Researcher**

A new study on patients who have undergone total laparoscopic hysterectomy surgery has been planned by the Department of Nursing, Hamidiye Institute of Health Sciences, University of Health Sciences. The name of the study is "The Effect of Chewing Gum on Intestinal Functions and Pain Level After Total Laparoscopic Hysterectomy Surgery".

Participation in the study is based on volunteerism. We would like to inform you about the research before your decision. After reading and understanding this information, if you want to participate in the research, please sign the form.

The reason we would like to do this research is to determine whether chewing gum after total laparoscopic hysterectomy operations has an effect on intestinal function and pain. Your participation in this study is important for the success of the research. Having undergone laparoscopic surgery of chewing gum

The above information about this research was conveyed to me by Mr. Senay Demirbaş Meydan stating that a medical research will be conducted at the Department of Nursing of Hamidiye Institute of Health Sciences of the University of Health Sciences. After this information, I was invited as a "participant" in such a study. If I participate in this study, I believe that the confidentiality of the information belonging to me that should remain between me and the researcher will be approached with great care and dec during this research. I was given enough confidence that my personal information would be protected by my application during the use of the research results for educational and scientific purposes. During the execution of the project, I can withdraw from the research without giving any reason. (However, I am aware that it would be appropriate for me to inform the researchers in advance that I will withdraw from the study so as not to leave them in a difficult situation) I can also be excluded from the research by the researcher provided that no harm is caused to my medical condition.

| The Participant | The Researcher Who Made the Statement |
|-----------------|----------------------------------------------|
| Name, Surname: | First Name, Last Name: Şenay Demirbaş Meydan |
| Address: | Tel: 0546 924 91 04 |
| | Signature: |
| Tel: | Date: |
| Signature: | |
| Date: | |

## INFORMED VOLUNTARY REGISTRATION FORM (CONTROL GROUP)

### **Dear Participant**

A new study on patients who have undergone total laparoscopic hysterectomy surgery has been planned by the Department of Nursing, Hamidiye Institute of Health Sciences, University of Health Sciences. The name of the study is "The Effect of Chewing Gum on Intestinal Functions and Pain Level After Total Laparoscopic Hysterectomy Surgery".

Participation in the study is based on volunteerism. We would like to inform you about the research before your decision. After reading and understanding this information, if you want to participate in the research, please sign the form.

The reason why this research is wanted is to determine whether chewing gum after total laparoscopic hysterectomy operations has an effect on intestinal functions and pain. Your participation in this study is important for the success of the research. If you agree to participate in the study, you can apply at the clinic

The above information about this research was conveyed to me by Mr. Senay Demirbaş Meydan stating that a medical research will be conducted at the Department of Nursing of Hamidiye Institute of Health Sciences of the University of Health Sciences. After this information, I was invited as a "participant" in such a study. If I participate in this study, I believe that the confidentiality of the information belonging to me that should remain between me and the researcher will be approached with great care and dec during this research. I was given enough confidence that my personal information would be protected by my application during the use of the research results for educational and scientific purposes.

During the execution of the project, I can withdraw from the research without giving any reason. (However, I am aware that it would be appropriate for me to inform the researchers in advance that I will withdraw from the study so as not to leave them in a difficult situation) I can also be excluded from the research by the researcher provided that no harm is caused to my medical condition.

| The Participant | The Researcher Who Made the Statement |
|-----------------|----------------------------------------------|
| Name, Surname: | First Name, Last Name: Şenay Demirbaş Meydan |
| Address: | Tel: 0546 924 91 04 |
| | Signature: |
| Wire: | History: |
| Signature: | |
| History: | |